CLINICAL TRIAL: NCT04315571
Title: Effective Ascites ReLief In earlY TIPS (EARLY TIPS) Using Viatorr CX vs. LVP Study
Brief Title: Comparing Ascites Relief In Two Standard Treatments: Large Volume Paracentesis Vs. Early Tips Using Viatorr Controlled Expansion Stents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: W.L.Gore & Associates (Industry)
Responsible Party: Principal Investigator, Edward Wolfgang Lee, MD, Associate Professor of Radiology and Surgery, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CXTIPSvLVP-v1
Record Dates: First submitted 2020-03-09; First posted 2020-03-19 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hypertension, Portal; Ascites
Keywords: end-stage liver disease; hepatic encephalopathy; cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Ascites; End Stage Liver Disease; Hepatic Encephalopathy; Fibrosis | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Routine Large Volume Paracentesis (LVP) with albumin infusion
  Interventions: Procedure: Large Volume Paracentesis with albumin infusion
- Group B (Active Comparator): Early Transjugular intrahepatic portosystemic shunt (TIPS) procedure using Gore Viatorr CX
  Interventions: Device: Gore® Viatorr® Endoprosthesis with controlled expansion

INTERVENTIONS:
Device: Gore® Viatorr® Endoprosthesis with controlled expansion — TIPS (Transjugular Intrahepatic Portosystemic Shunt) is a minimally invasive procedure in which a new path is made through the liver to carry blood from the portal vein to the heart, thus helping to alleviate the problems associated with elevated portal vein pressure.
  Other Names: TIPS
  Arms: Group B
Procedure: Large Volume Paracentesis with albumin infusion — For therapeutic (large-volume) paracentesis, a 14-gauge cannula attached to a vacuum aspiration system is used to collect up to 8 L of ascitic fluid. Concurrent infusion of IV albumin is recommended during large-volume paracentesis to help avoid significant intravascular volume shift and postprocedural hypotension.
  Other Names: LVP with albumin infusion
  Arms: Group A

SUMMARY:
For this study, the investigators will be collecting data based on patients' random selection to two different approved standard of care treatments for ascites: Subjects will get randomized into either Group A: Large Volume Paracentesis (LVP) with albumin infusion, or Group B: an early transjugular intrahepatic portosystemic shunt (TIPS) procedure.

DETAILED DESCRIPTION:
End Stage Liver Disease (ESLD) severely impacts body function leading to elevated blood pressure within the liver called "portal hypertension." One of its subsequent symptoms is ascites, or fluid accumulation in the abdomen. One standard treatment to relieve ascites is large volume paracentesis (puncture of the abdomen to drain the fluid). Another standard treatment is the TIPS procedure, which involves creating a shunt (small passage allowing fluid movement) within the liver to relieve the increased blood pressure in the liver.

For this study, the investigators will be collecting data based on patients' random selection to two different approved standard of care treatments for ascites: Subjects will get randomized into either Group A: Large Volume Paracentesis (LVP) with albumin infusion, or Group B: an early transjugular intrahepatic portosystemic shunt (TIPS) procedure.

The study will include about 68 patients (34 patients will be selected for Group A: continuing conservative treatment of LVP with albumin infusion, and 34 patients will be selected for Group B: undergoing early TIPS with Gore®Viatorr®CX). Each patient will be followed up at 1 month, 3 months, 6 months, and 12 months.

The primary objective of this study is to evaluate the overall clinical efficacy in symptom relief of ascites of patients receiving the Gore® Viatorr® CX in early TIPS procedures compared to LVP (large volume paracenthesis). In order to so, the investigators will be using information found in patient medical records, collected as a part of standard of care, to analyze clinical outcomes, complications, and the rate of secondary interventions at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Males and females > 18 years of age at time of procedure
* First de novo TIPS placement
* Patent internal or external jugular vein
* Willing to provide the hepatology service information for follow up
* No known diagnosis of hypercoagulopathy
* No portal vein thrombosis
* No malignancy (must be a definite diagnosis)
* Patient must provide written informed consent
* Proper clinical indication of TIPS based on American Association for the Study of Liver Diseases (AASLD) guidelines

  * Recurrent ascites necessitating at least 2 large volume paracenteses performed within a minimum interval of 3 weeks

Exclusion Criteria:

* Age <18
* LVP > 6 times in 2 months
* Liver failure (Child Pugh > 12)
* Cardiac failure
* No right jugular venous access
* Absolute TIPS contraindications (e.g. right heart failure, severe encephalopathy, liver failure, pregnant (if possible)).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of Paracentesis | 1 year post-procedure
  The average number of paracentesis per week.

SECONDARY OUTCOMES:
Transplant free survival | 1 year post-procedure or until the patient expires or receives transplant
  Overall survival without transplant after the treatment

OTHER OUTCOMES:
Stent diameter change | 1 month and 6 months
  Stent diameter changes from the time of TIPS placement

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Lee, MD, PhD, Principal Investigator — University of California
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Velasco Hidalgo L, Flores Garcia NC, Aguirre-Salgado MI. Transjugular intrahepatic portosystemic shunts for adults with hepatorenal syndrome. Cochrane Database Syst Rev. 2024 Jan 18;1(1):CD011039. doi: 10.1002/14651858.CD011039.pub2. PMID 38235907